CLINICAL TRIAL: NCT02248493
Title: The Effect of Intravenous Paracetamol in Combination With NSAIDs for Postoperative Pain in Children
Brief Title: Intravenous Paracetamol for Postoperative Pain
Acronym: IVPARACET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Danguole C Rugyte, MD, PhD, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BEC-MF-10
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Pain, Postoperative; Recovery of Function; Child
Keywords: Pain, Postoperative; Paracetamol; Administration, Intravenous; Anti-Inflammatory Agents, Non-Steroidal; Child; Adolescent
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Saline Solution; Ketoprofen; Tramadol; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- paracetamol and ketoprofen (Experimental): paracetamol 20 mg/kg (1% 2 ml/kg) IV at the end of surgery 6 and 20 hours thereafter.
  ketoprofen 1.5 mg/kg IV at the end of surgery 8 and 16 hours thereafter. tramadol 2 mg/kg IV on patient request up til 4 mg/kg or PCA morphine during 24 hours postoperatively.
  Interventions: Drug: Paracetamol; Drug: Ketoprofen; Drug: Tramadol; Drug: Morphine
- placebo and ketoprofen (Placebo Comparator): 0.9% sodium chloride (2 ml/kg) IV at the end of surgery 6 and 20 hours thereafter.
  ketoprofen 1.5 mg/kg IV at the end of surgery 8 and 16 hours thereafter. tramadol 2 mg/kg IV on patient request up til 4 mg/kg or PCA morphine during 24 hours postoperatively.
  Interventions: Drug: Placebo (for paracetamol); Drug: Ketoprofen; Drug: Tramadol; Drug: Morphine

INTERVENTIONS:
Drug: Paracetamol
  Other Names: Acetaminophen
  Arms: paracetamol and ketoprofen
Drug: Placebo (for paracetamol)
  Other Names: 0.9% sodium cloride solution; Normal saline solution; Izotonic saline solution
  Arms: placebo and ketoprofen
Drug: Ketoprofen
  Other Names: Ketonal
Drug: Tramadol — Administered on request as rescue medication in a dose 2 mg/kg IV up till 2 doses. No other opioid is given to these patients.
  Other Names: Tramal
Drug: Morphine — administered in patients receiving IV PCA with morphine postoperatively. No other opioid is given to these patients.

SUMMARY:
The purpose of this study is to define if intravenous paracetamol may improve analgesia and outcome in pediatric surgical patients treated with non-steroidal anti-inflammatory drugs (NSAIDs) postoperatively.

Hypothesis: intravenous paracetamol in a dose 60 mg/kg/24 h IV, given in addition to IV ketoprofen (4,5 mg/kg/24h), improves analgesia and physical recovery in children and adolescents following surgery.

DETAILED DESCRIPTION:
Patients aged 1-18 years undergoing general, plastic or orthopedic surgery with expected moderate to severe pain at least for 24 hours postoperatively, who meet inclusion criteria and does not meet exclusion criteria, are enrolled. At the end of surgical procedure, at skin closure, all patients are given 1,5 mg/kg intravenous ketoprofen and repeated every 8 hours up till 4,5 mg/kg/24 h. Patients in paracetamol group are additionally given the first dose of IV paracetamol 20 mg/kg and repeated 6 and 20 hours postoperatively up till 60 mg/kg/24 h. Patients in the placebo group are given 0.9% sodium chloride 2 ml/kg IV and repeated 6 and 20 hours postoperatively.

After surgery optional rescue analgesia is given on patient request: either tramadol in a dose of 2 mg/kg (up till 4 mg/kg/24h), either patient-controlled analgesia (PCA) with morphine, as indicated according to the standard of care. Patients are evaluated up till 24 hours postoperatively. After that patients are followed up as long as indicated per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients 1-18 years of age, undergoing general, plastic or orthopedic surgery with expected median to severe pain postoperatively.
* physical status of the patient corresponding to American Society of Anesthesiologists (ASA) class 1 or 2
* Signed written informed consent by parents/official caregivers.

Exclusion Criteria:

* Allergy to paracetamol, ketoprofen, tramadol, morphine or any NSAID
* oncologic disease
* central nervous system disease
* renal dysfunction
* hepatic dysfunction
* bronchial asthma
* ulcer(s) in gastrointestinal system
* hemorrhagic diathesis
* chronic use of NSAIDs
* chronic use of opioids
* chronic use of anticoagulants
* female patient is known to be pregnant

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2012-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
change in postoperative intravenous opioid dose | 24 hours postoperatively

SECONDARY OUTCOMES:
change in pain level (analgesia) assessed by 10 point pain scales | 1 hour postoperatively
change in pain level (analgesia) assessed by 10 point pain scales | 24 hours postoperatively

OTHER OUTCOMES:
time until the first oral intake after surgery | 24 hours postoperatively
time until the first urination after surgery | 24 hours postoperatively
time until ambulation after surgery | 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Danguole C Rugyte, MD. PhD, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Lithuanian University of Health Sciences Kaunas Clinics, Kaunas, Lithuania

REFERENCES:
- [Background] Ong CK, Seymour RA, Lirk P, Merry AF. Combining paracetamol (acetaminophen) with nonsteroidal antiinflammatory drugs: a qualitative systematic review of analgesic efficacy for acute postoperative pain. Anesth Analg. 2010 Apr 1;110(4):1170-9. doi: 10.1213/ANE.0b013e3181cf9281. Epub 2010 Feb 8. PMID 20142348
- [Background] Wong I, St John-Green C, Walker SM. Opioid-sparing effects of perioperative paracetamol and nonsteroidal anti-inflammatory drugs (NSAIDs) in children. Paediatr Anaesth. 2013 Jun;23(6):475-95. doi: 10.1111/pan.12163. Epub 2013 Apr 9. PMID 23570544
- [Background] Hiller A, Silvanto M, Savolainen S, Tarkkila P. Propacetamol and diclofenac alone and in combination for analgesia after elective tonsillectomy. Acta Anaesthesiol Scand. 2004 Oct;48(9):1185-9. doi: 10.1111/j.1399-6576.2004.00473.x. PMID 15352967
- [Background] Rugyte D, Kokki H. Intravenous ketoprofen as an adjunct to patient-controlled analgesia morphine in adolescents with thoracic surgery: a placebo controlled double-blinded study. Eur J Pain. 2007 Aug;11(6):694-9. doi: 10.1016/j.ejpain.2006.11.001. Epub 2006 Dec 20. PMID 17185016